CLINICAL TRIAL: NCT04013204
Title: Endothelial Function Guided Therapy in Patients With Non-obstructive Coronary Artery Disease (EndoFIND Study)
Brief Title: Endothelial Function Guided Therapy in Patients With Non-obstructive Coronary Artery Disease
Acronym: EndoFIND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Mayo Clinic (Other); Peking University Shougang Hospital (Other)
Responsible Party: Principal Investigator, Wang Hongyu, Professor, Peking University Clinical Research Institute, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PUCRI-2019- EndoFIND-01
Record Dates: First submitted 2019-07-01; First posted 2019-07-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Non-obstructive Coronary Artery Disease
Keywords: non invasive endothelial function test; non-obstructive coronary artery disease; Major Adverse Cardiovascular Events

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, patient and assessor blinded, parallel control, two-stage, clinical trial.
  Phase I: a feasibility study to collect data on key process outcomes including physician's prescription behaviors, patients' cardiovascular risk, and trend of reduction in cardiovascular events, To create an initial and to inform for the Phase II larger multicenter trial on choosing clinical endpoints and sample size.
  Phase II: will extend all patients from Phase I to a longer period of follow up and recruit more new patients to enlarge the sample size, in order to have a full study on the effect of introducing EFT as a routine test in reducing clinical endpoint (major adverse cardiovascular events) among patients with NOCAD.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is patient and assessor blinded; that is, both groups of patients are unaware of the endothelial function results. This study will use blind methods for endpoint data collectors; that is, the data collectors will collect secondary prevention medication and cardiovascular event data for coronary artery disease without an awareness of patient grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: Before the patient returns to the doctor and the prescription is issued, the EDCM system will feed back the EndoPAT test results to the responsible doctor through the automatically generated information on the doctor's mobile phone, but will not let the patient know the endothelium test results (blinded to the patient).
  Interventions: Other: Endothelial function guided therapy
- Control group (No Intervention): Control group: The EDCM system will not report the EndoPAT test results to the responsible doctor (the doctor cannot see the final EFT results), nor can the patients know the EFT results.

INTERVENTIONS:
Other: Endothelial function guided therapy — To evaluate the effect of integration of non invasive endothelial function test (EFT) as a routine test in increasing appropriate treatment to reduce cardiovascular risk including prescription of lipid, blood pressure and glucose lowering medications by physicians at the clinic for patients with non-obstructive coronary artery disease (NOCAD) and the effect of introducing EFT as a routine test in reducing clinical endpoint (major adverse cardiovascular events) among patients with non-obstructive coronary artery disease(NOCAD).
  Arms: Intervention group

SUMMARY:
The purpose of this study is to systematically evaluate the clinical application value of vascular endothelial function examination in patients with non-obstructive coronary artery disease.

DETAILED DESCRIPTION:
The study will be carried out in two stages. Phase I is mainly intended to evaluate the effects of vascular EFT on the prescription of doctors and the application rate of mid and long-term secondary prevention medication in patients. If the results are positive, the sample size and observation time will be further expanded in Phase II to evaluate its impact on the cardiovascular events of patients, as well as its cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 years or older;
* 2. Patients with NOCAD defined by CT or CAG results of less than 50% occlusion;
* 3. Having signed their written informed consent.

Exclusion Criteria:

* 1. Left ventricular ejection fraction ≤ 50%;
* 2. Serious endocrine diseases (severe hyperthyroidism, hypothyroidism);
* 3. Severe liver diseases (jaundice hepatitis, liver cirrhosis, liver failure);
* 4. Severe nephropathy (uremia, renal failure);
* 5. Severe inflammatory diseases (severe infection, lupus erythematosus, etc.);
* 6. Malignant tumor;
* 7. Mental disorders or cognitive disorders;
* 8. Participating in other interventional clinical trials;
* 9. There are any other factors that the treating doctors think are not suitable for inclusion or completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Compliance rate of patients to physicians prescription | up to 30 months
  The incidence number of patients compliance to guidelines based medical therapy with prescription of cholesterol, blood pressure and glucose lowering medications by physicians at clinic for patients with non-obstructive coronary artery disease.
Total incidence number of Major Adverse Cardiovascular Events | up to 54 months
  The incidence number of MACE(Major Adverse Cardiovascular Events) including total death, non-fatal AMI or stroke(including stroke revascularization).

SECONDARY OUTCOMES:
Mean improvement of endothelial function | up to 30 months
  The mean improvement in endothelial function from baseline to 12 months, estimated by RHI(Reactive Hyperemia Index).
Incidence number of Major Adverse Cardiovascular Events | up to 30 months
  The incidence number of MACE(Major Adverse Cardiovascular Events) during 0 to 12 months
Reduction of lipid levels | up to 30 months
  The reduction in lipid levels from baseline to 12 months
Reduction of blood pressure | up to 30 months
  The reduction in blood pressure from baseline to 12 months
Compliance rate of patients with treatment target | up to 30 months
  The percentage of patients with treatment target attained in terms of hypertension, diabetes, and dyslipidemia at 12 months after baseline.
Compliance rate of patients with appropriate prescription by physicians | up to 30 months
  The percentage of patients with appropriate prescription of cholesterol, blood pressure and glucose lowering medications by physicians at 3, 6 and 12 months after baseline.
Compliance rate of patients with healthy life style | up to 30 months
  The percentage of patients with healthy life style at 3, 6 and 12 months after baseline. The healthy life style is defined as having no smoking, physical activities with at least 3 times a week and 30 min per time, BMI<25 Kg/M2.
Cost-effectiveness rate of Endothelial Function Testing | up to 54 months
  The cost-effectiveness incremental ratio of Endothelial Function Testing in reducing MACE(Major Adverse Cardiovascular Events) .

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Wang, MD, Principal Investigator — Peking University; Gaoqiang Xie, PHD, Study Director — Peking University
Locations (1):
- Peking University Shougang Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hwang IC, Jeon JY, Kim Y, Kim HM, Yoon YE, Lee SP, Kim HK, Sohn DW, Sung J, Kim YJ. Association between Aspirin Therapy and Clinical Outcomes in Patients with Non-Obstructive Coronary Artery Disease: A Cohort Study. PLoS One. 2015 Jun 2;10(6):e0129584. doi: 10.1371/journal.pone.0129584. eCollection 2015. PMID 26035823